CLINICAL TRIAL: NCT01977417
Title: Inflammation Inhibition for Microvascular and Autonomic Dysfunction in Obese Prediabetic Humans
Brief Title: Inflammation Inhibition in Prediabetic Humans
Acronym: INCITE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Gary L. Pierce (Other)
Responsible Party: Sponsor-Investigator, Gary L. Pierce, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201209707
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Prediabetes; Obese
Keywords: Endothelial Function; Arterial Stiffness; Inflammation; Muscle Sympathetic Nervous System; Prediabetes; Autonomic function
MeSH Terms: conditions — Prediabetic State; Obesity; Inflammation | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Salsalate (Experimental): 3.0 grams/day salsalate (1.5 g twice per day)
  Interventions: Drug: Salsalate
- Placebo (Placebo Comparator): Placebo capsule twice per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salsalate
  Arms: Salsalate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Prediabetes, characterized by elevated fasting blood sugar or exaggerated blood sugar response to sugar ingestion, effects over 79 million adult Americans and is a precursor to the development of Type 2 diabetes. Importantly, approximately 42% of Iowans (950,000) have diabetes and 32% (670,000) have prediabetes with the majority of those with prediabetes going undiagnosed. Adults with prediabetes demonstrate early signs of cardiovascular and nervous system abnormalities and are at high risk for developing overt diabetes unless aggressive lifestyle (weight loss, exercise) or pharmacological interventions are employed. Interestingly, data in recent years has linked obesity and diabetes to chronic inflammation of the blood vessels and brain areas that regulate blood pressure. Therefore, the current study will test whether a commonly used aspirin-like anti-inflammatory drug called salsalate, will improve blood vessel health and nervous system dysfunction in adults with prediabetes. Eligible subjects will have measurements of blood pressure, blood vessel function in the arms and eyes, assessments of nerve activity, and blood samples taken before and after 4 weeks of ingesting an FDA approved aspirin-like drug called salsalate. The study is important because it will identify a potentially new pharmacological strategy to treat vascular and nervous system abnormalities in overweight and obese adults with early stage type 2 diabetes using an inexpensive, generically available drug with an excellent safety record that has been used for decades to treat chronic inflammatory conditions such as rheumatoid arthritis. If proven effective, this will provide preliminary support for the concept of targeting inflammation as a new clinical approach to treating early diabetes related complications. Furthermore, the current pilot study will provide support for developing a larger clinical trial using salsalate that could potentially then be extended to patients with type 2 diabetes and cardiovascular disease, as well as lead to the development of new anti-inflammatory agents with greater specificity for selective inflammatory pathways.

DETAILED DESCRIPTION:
A total of 30 healthy men and women ages 18-79 years who are obese defined as body mass index (BMI) of 30 kg/m2 or greater and with prediabetes (defined as fasting blood glucose between 100-126 mg/dl, a fasting blood glucose of 140-199 mg/dl at 120 min during an oral glucose tolerance test; or HbA1C of 6-6.5%) will be enrolled and randomized to 4-5 weeks of salsalate or placebo in the study. CONTROL GROUP: Another n=10 healthy obese men and women age 18-49 WITHOUT prediabetes will be enrolled for baseline testing but will not undergo randomization to the salsalate/placebo intervention. Therefore, total enrollment will be n=40.

All subjects will have no history of cardiovascular, metabolic or pulmonary disease as determined from medical history and physical exam, and a resting 12-lead ECG. Subjects may be on anti-hypertensive medications but will be asked to hold the medication on the morning of testing. Subjects on medications for Type I or II diabetes mellitus or for hyperlipidemia will be excluded (see complete list below). Subjects will be non-smokers or quit smoking at least one year ago. Women will have regular menses and will be tested during the early follicular phase of their menstrual cycle (within 8 days of onset of menses) to control for differences in circulating estradiol concentrations. Aim 1 will measure microvascular function and aortic wall stiffness in obese prediabetic adults before and after 1 month of salsalate or placebo. Hypothesis 1 is that chronic inflammation inhibition will improve microvascular and large elastic artery function in obese adults with prediabetes. Aim 2 will measure muscle sympathetic nervous system activity (MSNA) and baroreflex sensitivity in obese prediabetic adults before and after 1 month of salsalate or placebo. Hypothesis 2 is that chronic inflammation inhibition will decrease MSNA and improve baroreflex sensitivity in obese adults with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.

  * Age is > or = 18 and < or = 49 years (older)
  * Obese defined as body mass index > or = 30 kg/m2
  * Prediabetic defined as fasting blood glucose 100-126 mg/dl, blood glucose between 140-199 mg/dl at 120 min of oral glucose tolerance test
  * healthy, as determined by health history questionnaire, medical history and physical examination by physician or nurse practitioner, blood chemistries, resting blood pressure and exercise 12-lead ECG
  * blood chemistries indicative of normal renal function (creatinine <2.2 mg/dl), liver (<3 times upper limit for ALT, AST), and thyroid function (TSH between 0.4 - 5.0 mU/L)
  * If currently receiving treatment with or taking any of the following supplements, be willing and able to discontinue taking them for 2 weeks prior and throughout the treatment period: Vitamin C, E or other multivitamins containing vitamin C or E; nutraceuticals containing vitamin C or E
  * No history of cardiovascular disease (e.g., heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy), Type 1 or 2 diabetes mellitus, or peripheral arterial disease
  * Sedentary or recreationally active defined as performs regular aerobic exercise (30 min or more of vigorous walking, jogging, swimming, cycling, etc) less than 2 days/week or less than 12 days/month over the last year
  * Non-smokers, defined as no history of smoking, no smoking for at least the past 1 year
  * Normal resting 12-lead ECG.

Exclusion Criteria:

* History of cardiovascular disease such as myocardial infarction, stroke, heart failure with or without LV ejection fraction <40%, cardiomyopathy, valvular heart disease, cardiomyopathy, heart transplantation, Type 2 diabetes and Type 1 diabetes

  * Smoking or history of smoking within past one year
  * History of gastric ulcers, bleeding disorders, dyspepsia, severe gastroesophageal reflux disease (GERD), or metabolic acidosis
  * History of asthma or lung disease (chronic obstructive pulomonary disease, COPD)
  * Abnormal resting 12-lead ECG (e.g., evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter)
  * Serious neurologic disorders including seizures
  * History of renal failure, dialysis or kidney transplant
  * Serum creatinine > 2.2 mg/dL, or hepatic enzyme concentrations > 3 times the upper limit of normal
  * History of HIV infection, hepatic cirrhosis, other preexisting liver disease, or positive HIV, Hepatitis B or C test at screening.
  * Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
  * History of recent chicken pox, shingles or influenza (ie., risk of Reye's syndrome) Recent flu-like symptoms within the past 2 weeks
  * Pregnant or breastfeeding at screening, or planning to become pregnant (self or partner) at any time during the study. A urinary pregnancy test will be done on all females. If test is positive, the subject will be excluded.
  * Women with history of hormone replacement therapy within the past 6 months
  * History of rheumatoid arthritis, Grave's disease, systemic lupus erythamatosis, and Wegener's granulomatosis;
  * Taking medications for diabetes mellitus, kidney disease, liver disease, asthma, sepsis or seizure disorders;
  * Taking lipid lowering (e.g., statins, niacin), glycemic control (e.g. metformin, insulin), anticoagulation, anti-seizure, anti-depression or antipsychotic agents
  * History of co-morbid condition that would limit life expectancy to < 6 months.
  * It is unknown if Salsalate is transferred in seminal fluid of men. However, it is recommended that proper protection such as a condom be used during intercourse during the study.
  * Concomitant treatment with: aspirin, baby aspirin, indomethacin, naproxen (Aleve), acetaminophen (Tylenol), ibuprofen (Advil, Motrin), any other non-steroidal anti-inflammatory drugs; cox-2 inhibitors (Celebrex, Vioxx, etc); allopurinol (Zyloprim, Lopurin, Alopurin; coumadin (Wafarin), enoxaparin (Lovenox); clopidogrel (Plavix); dypyridamole (Persantine); heparin; diabetic medications (Metformin, glyburide, insulin, etc), TZDs (Avandia, Rezulin, Actos); corticosteroids (prednisone); methotrexate, infliximib (Remicade), etaneracept (Enbrel); levothyroxine (Levoxyl, Synthroid, Levoxyl, Unithroid); Levodopa; Phosphodiesterase (PDE) 5 inhibitors (e.g., Viagra®, Cialis®, Levitra®, or Revatio®); PDE 3 inhibitors (e.g., cilostazol, milrinone, or vesnarinone); lithium
  * May participate if use of the following medications are discontinued 2 weeks prior to participation: salicylate medications, aspirin, antioxidants, herbal supplements, vitamins, omega-3 fatty acids; cox-2 inhibitors (Celebrex, Vioxx, etc)
  * May participate if no use of the following medications in the 48 hours prior to experimental visits: naproxen (Aleve), acetaminophen (Tylenol), ibuprofen (Advil, Motrin), other any non-steroidal anti-inflammatory drugs
  * Vulnerable populations (prisoners, etc.) are not included in this study because we are studying healthy middle-aged/older adults.
  * Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
  * Hemoglobin <12 mg/dl for men; < 10 mg/dl for women
  * History of alcohol abuse or >10 alcoholic units per week (1 unit= 1 beer, 1 glass of wine, 1 mixed cocktail containing 1 oz alcohol)
  * Low platelets (<100,000 cu mm)
  * On weight loss drugs (e.g., Xenical (orilistat), Meridia (sibutramine), Acutrim (phenylpropanol-amine), or similar over-the-counter medications) within 3 months of screening
  * Any surgery within 30 days of screening

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Pierce, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Salsalate: 3.0 grams/day salsalate (1.5 g twice per day)
  Salsalate
- Placebo: Placebo capsule twice per day
  Placebo
Period: Overall Study
Arm/Group | Salsalate | Placebo
Started | 8 | 13
Completed | 5 | 7
Not Completed | 3 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Female enrollment goal met | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salsalate | Placebo | Total
Number analyzed (Participants) | 8 | 13 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (15.7) | 28.1 (10.0) | 31.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 13 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: Vascular Endothelial Function in Obese Prediabetic Adults Before and After 1 Month of Salsalate or Placebo.
Description: Brachial artery flow-mediated dilation
Time Frame: Change from baseline at 4 weeks
Measure: Mean (Standard Deviation); unit: % dilation
Arm/Group | Salsalate | Placebo
Number analyzed (Participants) | 5 | 7
% dilation | 5.57 (4.35) | 6.98 (6.43)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Participant called in on day 4 and reported they developed punctate rash on bilaterally around wrists and ankles that was itching and red blotchy, but no facial swelling, no trouble breathing or swallowing, no wheezing. Participant was evaluated by study physician over the phone and was instructed to stop medication and then examined in the clinical research unit on day 6 and reported the rash had decreased since day 4 and the rash resolved completely within a few days.
Arm/Group | Salsalate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/13
Other Adverse Events (participants affected / at risk) | 1/8 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Salsalate (N=8) | Placebo (N=13)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT01977417/Prot_SAP_000.pdf